CLINICAL TRIAL: NCT02041884
Title: Psychological Treatment Through Internet and Smartphones for Adults With Attention Deficit Hyperactive Disorder (ADHD) - a Randomized Controlled Trial
Brief Title: CBT Through Internet and Smartphones for Adults With ADHD - a Randomized Controlled Trial
Acronym: Ad5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/333-31
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: ADHD
Keywords: Cognitive Behavioral Therapy; Dialectical Behavioral Therapy; Applied Relaxation; Stress-reduction; Smartphone application; ADHD; Randomized controlled trial; Psychological treatment; Efficacy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- iCBT (Experimental): A skill training internet-based treatment program based on CBT and DBT interventions .
  Interventions: Behavioral: iCBT for Adults with ADHD
- Internet stress-reduction (Active Comparator): Internet-based psychoeducation, stress-reduction, and Applied Relaxation based on CBT (control group)
  Interventions: Behavioral: Internet stress-reduction
- Treatment as usual (TAU)/waiting list (Other): Treatment as usual (usually medications for ADHD), will be offered treatment after the FU3 (week 24)
  Interventions: Other: Treatment as usual (TAU)/waiting list

INTERVENTIONS:
Behavioral: iCBT for Adults with ADHD — A skill training internet-based treatment program based on CBT and DBT interventions .
  Arms: iCBT
Behavioral: Internet stress-reduction — Internet-based psychoeducation, stress-reduction, and Applied Relaxation based on CBT (control group)
  Arms: Internet stress-reduction
Other: Treatment as usual (TAU)/waiting list — Treatment as usual (usually medications for ADHD), will be offered treatment after the FU3 (week 24)
  Arms: Treatment as usual (TAU)/waiting list

SUMMARY:
The purpose of this study is to further evaluate the treatment for adults with ADHD used in our previous study (clinicaltrials.gov ID NCT01659164). It will now be converted to therapist supported, internet-delivered cognitive behavioral therapy (iCBT) with an additional smartphone application and evaluated through a randomized controlled trial during 12 weeks. The patients will be randomized to one of three conditions

* an active treatment group where the intervention is based on cognitive - and dialectical behavioral therapy (CBT and DBT) and the mobile app.
* an active ICBT-treatment based on psychoeducation, a CBT stress-reduction program and Applied Relaxation, and
* treatment as usual (TAU) / waiting list.

The main objective of the study is to evaluate if both of the treatment conditions will show better outcomes than TAU regarding decreased ADHD symptoms and increased functioning and life quality.

Another objective is to evaluate if the group receiving the active iCBT treatment (based on CBT and DBT) will show better outcomes in comparison to the control group regarding ADHD symptoms, overall functioning and life quality.

DETAILED DESCRIPTION:
Approximately one-third of children with ADHD continue to be fully symptomatic into adulthood and many of the remainders often retain some residual problems that require treatment. Thus ADHD is a prevalent and chronic disabling disorder. Drugs provide first line treatment for adults with ADHD but are not enough for everybody, while we still lack proper evidence for promising psychological treatment. In addition to core symptoms of ADHD including regulatory difficulties of attention, activity level and impulses, difficulties with emotional regulation are common.

Follow-up studies of adults with ADHD have shown that only a few patients were offered sufficient treatment and support after the neuropsychiatric assessment and testing. The majority of adults diagnosed with ADHD are offered pharmacological treatment (stimulant medication) as the sole treatment. However, stimulant medication is not effective for up to 20-50 percent of adults as they may not experience symptom reduction or they are unable to tolerate the medication.

Consequently, the possible benefits of identifying and treating individuals with ADHD are extensive. Treatment of ADHD is preferably multimodal, i.e. consisting of more than one intervention.

Although literature regarding psychological treatment is relatively limited, studies of cognitive behavioral therapy (CBT) and dialectical behavior therapy (DBT) show that structured short-term therapies are promising in reducing ADHD related symptoms and increasing life quality. The main treatment focus is to enhance executive and organizational skills, improvement of consequence thinking and impulse control as well as emotion regulation skills. However, the range of trained psychologist in this field is rather limited. Using internet for delivering evidence-based psychological treatment can therefore be a innovative treatment alternative in order to make inaccessible treatment available to a large group of patients with ADHD.

The actual treatment project aims to evaluate if adults with ADHD can benefit from psychological treatment delivered through Internet. About 150-200 patients will be recruited through several outpatient clinics in Stockholm. They will be randomized to one of three conditions - active psychological treatment (based on CBT and DBT), an active alternative treatment where they undergo a psychoeducational support program (based on CBT) or to treatment as usual (TAU) / waiting list. The patients in the treatment conditions will have a personal contact via the internet with a psychologist within the 12 week treatment period. Assessments will be done before, during and after treatment, and after 3 and 12 months. The patients in the TAU condition will be offered iCBT treatment after they have filled out the post assessments (after 12 weeks and at 3rd month after treatment).

ELIGIBILITY:
Inclusion Criteria:

* Swedish citizen
* Clinical diagnosis of AD/HD according to DSM-IV or DSM-5
* Age 18-65
* 17 or more on the Adult ADHD Self Report Scale (ASRS v1.1)
* Not medically treated for adhd symptoms, or medically treated with central stimulants or comparable substance since at least one month with no significant changes in dosage and where no change in medical treatment is anticipated during the study time frame for the participant. No change in any other medical treatment is anticipated during the study time frame for the participant.
* Participant are by investigators considered able to follow through the training protocol and take part in measures taken during the study time frame
* The participant hasn´t used drugs the last 3 months
* Access to, and ability to use the Internet and mobile phone during the study time
* ability to understand Swedish in speech and writing

Exclusion Criteria:

* Diagnosed substance abuse according to DSM-IV or DSM-5 criteria within 3 months prior to screening. Earlier episodic substance abuse is not excluding
* Co-existing psychiatric condition that investigators believe will unable the participant to follow through the training protocol and take part in measures taken during the study time frame.
* IQ ≤85 according to a neuropsychological assessment
* Suicidality risk which is assessed during the first assessment interview.
* Organic brain syndrome
* Serious somatic condition which will unable the participant to participate (through the training protocol)or, is anticipated to have a negative impact on the treatment results
* Autism spectrum disorder where the function level is deemed too low for the treatment to be carried out which is defined as moderate or severe problems scale (level 2 and 3) according to DSM-5
* Severe depression defined by >34 p on MADRS-S or by a clinician´s assessment
* Other current psychological treatment for AD/HD or previous participation in such a treatment that is deemed to interfere with the study design
* severe writing and reading disabilities
* dyslexia of such degree that it impedes participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in ASRS- v 1.1 | Baseline, at the end of week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and 11 in treatment, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  ADHD Self Report Scale (ASRS) (self rating)

SECONDARY OUTCOMES:
Change (from baseline) in ADHD Rating Scale | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  ADHD Rating Scale - assessed by an expert rater blind to Group allocation
Change (from baseline) in EQ-5D | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Euroqol - (self report) to measure general health and quality of life
Change (from baseline) in ISI | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Insomnia Severity Index - (self report) to measure insomnia symptoms
Change (from baseline) in PSS-4 | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Perceived Stress Scale - (self report) to measure level of stress in everyday life
Change (from baseline) in SDS | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Sheehan Disability Scale - (self report) to measure level of disability in everyday life
Change (from baseline) in MADRS-S | Baseline, at the end of week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and 11 in treatment, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Montgomery-Åsberg Depression Rating Scale - (self report) to measure level of depression
Change (from baseline) in DERS | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Difficulties of Emotion Regulation Scale - (self report)
Change (from baseline) in AaQoL | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Adult ADHD Quality of Life Measure - self report
Change (from baseline) in SWLS | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Satisfaction With Life Scale (self report) - measuring life quality. To evaluate the impact of the intervention on quality of Life, only the first three items in the scale will be used since the last two includes the whole Life-span and not just how Life quality is percived at the moment.
Change (from baseline) in WAI-1 | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Work Ability Index (self report - one item) - a self estimation of working ability
Changes (from baseline) in CGI-S | Baseline, 12 weeks (post), 24 weeks (FU3), and after 60 weeks (FU12)
  Clinical Global Impression - Severity scale - assessed by a blind expert rater - measuring symptom severity

OTHER OUTCOMES:
Treatment evaluation | during treatment and after 12 weeks of treatment (post)
  The investigators design own questions in order to evaluate how the participants have experienced the intervention regarding to knowledge, usage of the treatment methods and possible difficulties that they have experienced during treatment.
CGI-I | 12 weeks (post) and after 3 and 12 months (post)
  Clinical Global Impression - Improvement scale (rated by a clinician in order to detect level of improvement or worsening due to treatment)
TCS | Filled out by the patient at the 1st and 5th week of treatment
  Treatment Credibility Scale (self report)
*CSQ-8 | 12 weeks (post)
  Client Satisfaction Questionnaire-8 (self report) - in order to evaluate the treatment satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, PhD/Ass prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienheten, Psykiatri Sydväst, SLSO, Stockholm, Sweden

REFERENCES:
- See also: Information about the study — http://www.internetpsykiatri.se